CLINICAL TRIAL: NCT02627521
Title: Optimizing Timing of Coronary Artery Bypass Surgery in Patients Presenting With Acute Coronary Syndrome and Treated With Second Generation ADP Receptor Antagonist
Brief Title: Optimizing Timing of CABG in Patients Presenting With ACS and Treated With Ticagrelor
Acronym: CABG-TIME
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REB#13-287
Record Dates: First submitted 2015-12-03; First posted 2015-12-11 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRU Guided CABG (Experimental): Timing of CABG surgery within 24 hours of reaching a normalized platelet function (NPF). NPF defined as a PRU value >235 or a PRU value between >170 and <235 for two consecutive days as documented by VerifyNow assay.
  Interventions: Procedure: PRU guided CABG; Device: VerifyNow assay; Drug: Ticagrelor
- CABG per standard of care (Active Comparator): Timing of CABG per standard of care
  Interventions: Procedure: CABG per standard of care; Device: VerifyNow assay; Drug: Ticagrelor

INTERVENTIONS:
Procedure: PRU guided CABG — Coronary Artery Bypass Surgery
  Arms: PRU Guided CABG
Procedure: CABG per standard of care — Coronary Artery Bypass Surgery
  Arms: CABG per standard of care
Device: VerifyNow assay — Platelet reactivity Units by VerifyNow assay
Drug: Ticagrelor — Ticagrelor administration prior to randomization

SUMMARY:
The administration of Ticagrelor have demonstrated superiority to Clopidogrel in patients presenting with acute coronary syndrome (ACS) and remains a first line therapy as an adjunct to aspirin for patients admitted with ACS. The patient population treated with Ticagrelor at an early time point includes non ST elevation myocardial (NSTEMI) patients and those undergoing primary angioplasty for ST elevation myocardial infarction (STEMI). It is estimated that 10-15% of patients presenting with ACS have advanced coronary artery disease requiring Coronary Artery Bypass Surgery (CABG). The treatment guidelines recommend a delay of 5-7 days for CABG surgery in these patients for normalization of Ticagrelor induced platelet inhibition to reduce the risk of peri-operative bleeding. This delay may expose these high risk patients to adverse cardiac events while waiting for Ticagrelor effect to wean off. Furthermore, this empirical application of 5-7 day delay in all patients may be unnecessary due to the significant inter individual variability in response to Ticagrelor. There is limited data to determine the optimum timing of CABG surgery in ACS patients treated with Ticagrelor. The present study will determine the optimum timing of CABG in ACS patients treated with a loading and/or maintenance dose of Ticagrelor.

ELIGIBILITY:
Inclusion Criteria:

* Accepted for CABG surgery
* Treatment with Ticagrelor within 48 hours

Exclusion Criteria:

* Anticoagulation therapy
* Prior CABG.
* Active bleeding or at high risk of bleeding
* Severe liver or renal disease.
* Hypersensitivity to ticagrelor
* History of intracranial hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | up to 30 day
  The primary efficacy endpoint of the study is the total length of hospital stay (LOS) for CABG surgery between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Asim Cheema, MD, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided